CLINICAL TRIAL: NCT01073566
Title: The Effects of Finesse on Glycemic Control in Adults With Diabetes Using MDI: Finesse vs. Pen or Syringe and Vial as Bolus Prandial Insulin Device
Brief Title: Feasibility Study of Finesse for Bolus Prandial Insulin Dosing Compared to Multiple Daily Injections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Calibra Medical, Inc. (Industry)
Collaborators: Nancy Bohannon, MD, Med. Corp. (Unknown); Henry Ford Health System (Other); Northwestern University (Other); University of Texas Southwestern Medical Center (Other); International Diabetes Center at Park Nicollet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VP-00007
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Results first posted 2012-04-09 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus
Keywords: Autoimmune Diseases; Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders; Immune System Diseases; Insulin; Metabolic Diseases
MeSH Terms: conditions — Diabetes Mellitus; Autoimmune Diseases; Endocrine System Diseases; Glucose Metabolism Disorders; Immune System Diseases; Insulin Resistance; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Finesse (Experimental): Finesse Insulin Delivery Patch
  Interventions: Device: Finesse
- Usual injection device (Active Comparator): Pen/Syringe
  Interventions: Device: Pen/Syringe (Usual injection device)

INTERVENTIONS:
Device: Finesse — Finesse Insulin Delivery Patch
  Other Names: Insulin Bolus Patch
  Arms: Finesse
Device: Pen/Syringe (Usual injection device) — Pen/Syringe
  Other Names: Insulin pen; Insulin syringe; Insulin injection device
  Arms: Usual injection device

SUMMARY:
The purpose of this study is to evaluate that Finesse, for prandial insulin bolusing when used in conjunction with basal insulin, achieves equivalent glycemic control when compared to multiple daily injections and to evaluate its preference.

DETAILED DESCRIPTION:
The aim of this feasibility study is to compare efficacy, device satisfaction and quality of life (QOL) in people with type 1 or 2 diabetes delivering mealtime insulin using a novel insulin bolus-patch (Finesse™; Calibra Medical, Inc., Redwood City, CA) versus current devices that deliver bolus insulin (pen/syringe). All subjects injected their basal insulin using their current pen/syringe.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus on intensive insulin therapy

Exclusion Criteria:

* Insulin pump therapy
* Current use of NPH or regular insulin
* Severe hypoglycemic episodes in prior 6 months
* Unstable cardiac disease, hepatic, or renal function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President Clinical Affairs, Study Director — Calibra Medical, Inc.
Locations (5):
- United States (5):
  - California Pacific Medical Center, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Henry Ford Health System, Detroit, Michigan
  - International Diabetes Center at Park Nicollet, Minneapolis, Minnesota
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Result] Bohannon N, Bergenstal R, Cuddihy R, Kruger D, List S, Massaro E, Molitch M, Raskin P, Remtema H, Strowig S, Whitehouse F, Brunelle RL, Dreon D, Tan M. Comparison of a novel insulin bolus-patch with pen/syringe injection to deliver mealtime insulin for efficacy, preference, and quality of life in adults with diabetes: a randomized, crossover, multicenter study. Diabetes Technol Ther. 2011 Oct;13(10):1031-7. doi: 10.1089/dia.2011.0047. Epub 2011 Jul 6. PMID 21732797

RESULTS

PARTICIPANT FLOW:
Groups:
- Finesse Then Usual Injection Device: Subjects in this group first used Finesse Patch to deliver bolus insulin for 6 weeks then switched back to their usual pen/syringe to deliver bolus insulin for the final 6 weeks
- Usual Injection Device Then Finesse: Subjects in this group first used their usual pen/syringe to deliver bolus insulin for 6 weeks then switched to Finesse Patch to deliver bolus insulin for the final 6 weeks
Period: Period 1 (6 Weeks)
Arm/Group | Finesse Then Usual Injection Device | Usual Injection Device Then Finesse
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0
Period: Period 2 (6 Weeks)
Arm/Group | Finesse Then Usual Injection Device | Usual Injection Device Then Finesse
Started | 19 | 19
Completed | 18 | 19
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Finesse Then Usual Injection Device | Usual Injection Device Then Finesse | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (15.5) | 44.9 (15.3) | 47.3 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 11 | 14 | 25
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Mean Daily Blood Glucose
Description: Equivalence of Finesse to Usual Injection Device in Mean Daily Blood Glucose
Time Frame: 6 weeks
Population: Intent to treat
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Groups:
- Finesse: Bolus Patch
Arm/Group | Finesse | Usual Injection Device
Number analyzed (Participants) | 38 | 38
mmol/L | 8.61 (0.28) | 9.02 (0.26)
Statistical Analysis 1: Comparison: Finesse vs Usual Injection Device; A two-period, two-treatment crossover ANOVA model was used to compare devices for continuous measures; Test type: Non-Inferiority or Equivalence — Pre-study power calculations determined that 28 completed subjects provided 90% power to detect equivalence for the primary endpoint of MDBG of bolus-patch compared to pen/syringe using a 2-sided alpha level of 0.05, when the margin of equivalence for MDBG is 1.11 mmol/L, the true mean difference is 0.0, and the standard deviation of the differences is 1.72 mmol/L; p = 0.098, ANOVA; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.97 to 0.16], Standard Error of Mean 0.24 — Finesse versus usual injection device

2. Secondary Outcome: Glucose Profiles Per Day
Description: Standard deviation of 7 daily blood glucose values (3 pre-meal, 3 post-meal, and bedtime) for 3 days
Time Frame: 6 weeks
Population: Intent to Treat
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Finesse | Usual Injection Device
Number analyzed (Participants) | 38 | 38
mmol/L | 3.18 (0.18) | 3.63 (0.17)
Statistical Analysis 1: Comparison: Finesse vs Usual Injection Device; This was conducted at a 2-sided alpha level of 0.05 and confidence intervals (CI) were calculated at 95%, 2-sided. A two-period, two-treatment crossover ANOVA model was used to compare devices for continuous measures; Test type: Superiority or Other; p = 0.004, ANOVA; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.80 to -0.17], Standard Error of Mean 0.15 — Finesse versus usual injection device

3. Secondary Outcome: Insulin Delivery System Rating
Description: Subject satisfaction with insulin delivery was assessed by self-report on the validated Insulin Delivery System Rating Questionnaire. Scale is 0-100. Higher score is better.
Time Frame: 6 weeks
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Finesse | Usual Injection Device
Number analyzed (Participants) | 38 | 37
units on a scale | 82.9 (14.5) | 54.9 (17.5)
Statistical Analysis 1: Comparison: Finesse vs Usual Injection Device; Higher number is better. The answers were scored on a scale of 0-100 to standardize as described in the original papers; Test type: Superiority or Other; p < 0.001, McNemar

4. Secondary Outcome: Self-reported Hypoglycemic Episodes
Description: Severe hypoglycemia is defined as episodes in which the patient experienced coma, seizure, or suspected seizure or impairment sufficient to require the assistance of another person and either the blood glucose level is measured and found to be <50 mg/dl or the clinical manifestations were reversed by oral carbohydrate, subcutaneous glucagon, or intravenous glucose.
Time Frame: 6 weeks
Population: Intent to treat
Measure: Number; unit: episodes
Arm/Group | Finesse | Usual Injection Device
Number analyzed (Participants) | 38 | 38
episodes | 0 | 0

ADVERSE EVENTS:
Arm/Group | Finesse | Usual Injection Device
Serious Adverse Events (participants affected / at risk) | 1/38 | 1/38
Other Adverse Events (participants affected / at risk) | 8/38 | 9/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Finesse (N=38) | Usual Injection Device (N=38)
Acute Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Finesse (N=38) | Usual Injection Device (N=38)
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 1 (1) | 0/37 (0)
Tooth ache (Gastrointestinal disorders) | 0 (0) | 1/37 (1)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 2/37 (2)
Medical device site reaction (General disorders) | 1 (1) | 0/37 (0)
Acute pyelonephritis (Infections and infestations) | 1 (1) | 0/37 (0)
Flu (Infections and infestations) | 1 (1) | 0/37 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1/37 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 4/37 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 0/37 (0)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0/37 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1/37 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0/37 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0/37 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0/37 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0/37 (0)

LIMITATIONS AND CAVEATS:
The short duration of the study precludes comments on longer-term outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No